CLINICAL TRIAL: NCT05570890
Title: Immediate Effect of Electrical Noise Stimulation on Neuromuscular Adaptation During Single-Leg Stance in Healthy Young
Brief Title: Immediate Effect of Electrical Noise Stimulation on Neuromuscular Adaptation of Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: YM111060E
Record Dates: First submitted 2022-08-14; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-07

CONDITIONS: Balanced; Electroencephalography; Electromyography
Keywords: Center of pressure; Electroencephalography; Electromyography; H reflex; Electrical noise stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant
Masking Description: The stimulation intensity is set under the sensory threshold, therefore participants will be masked in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sham stimulation on stable surface (Experimental): The participant will not receive stimulation and will stand on flat ground.
  Interventions: Device: Sham stimulation
- Noise stimulation on stable surface (Experimental): The participant will receive stimulation with intensity set at 90% of their sensory threshold and will stand on flat ground.
  Interventions: Device: electrical noise stimulation
- Sham stimulation on unstable surface (Experimental): The participant will not receive stimulation and will stand on foam.
  Interventions: Device: Sham stimulation; Device: Foam
- Noise stimulation on unstable surface (Experimental): The participant will receive stimulation with intensity set at 90% of their sensory threshold and will stand on foam.
  Interventions: Device: electrical noise stimulation; Device: Foam

INTERVENTIONS:
Device: electrical noise stimulation — The intensity of electrical noise stimulation will be set at 90% of the sensory threshold of each participant.
  Arms: Noise stimulation on stable surface; Noise stimulation on unstable surface
Device: Sham stimulation — Participants will not receive stimulation.
  Arms: Sham stimulation on stable surface; Sham stimulation on unstable surface
Device: Foam — The foam will be used to make an unstable surface.
  Arms: Noise stimulation on unstable surface; Sham stimulation on unstable surface

SUMMARY:
Noise stimulation had an immediate effect on improving balance control. The present study aimed to clarify the immediate neuromuscular adaptation induced by noise stimulation and find the correlation between neuromuscular adaptation and functional performance.

DETAILED DESCRIPTION:
The mechanism behind noise stimulation is called Stochastic Resonance which improves the detectivity of sensory input with the presence of noise, making sub-sensory threshold input detectable. Noise stimulation had been proved to improve postural control, Ia afferent sensitivity, and muscle activity of the tibialis anterior. With this evidence of the effect of noise stimulation on balance enhancement, the neuromuscular adaptation induced by noise stimulation has not been researched yet. Therefore, the present study aims to clarify the immediate effect of noise on neuromuscular regulation during postural control.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 40 years old
* without ankle injury history in 1 year
* without musculoskeletal or neurological diseases that would affect balance performance
* without visual impairment (except vision correction or no visual problems)
* without vestibular impairment.

Exclusion Criteria:

* subject who cannot tolerate the cutaneous electrical stimulation to induce H reflex
* single-leg stance (SLS) without support is shorter than 80 secs

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean sway path of the center of pressure | 40 seconds under each condition
  The mean sway path in mm will represent balance performance
Mean sway velocity of the center of pressure | 40 seconds under each condition
  The mean sway velocity in mm/sec will represent balance performance
Cortical excitability | 40 seconds under each condition
  Power spectrum density of EEG will calculated for representing cortical excitability.
Spinal reflex excitability | 40 seconds under each condition
  H reflex amplitude will represent the excitability of peripheral control from spinal level nerve system.
Co-activation index | 40 seconds after each condition
  Co-activation index will be calculated by EMG activity of Tibialis Anterior and Soleus muscle to represent the muscle activity.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Study Director — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The informed Consent Form used in this research does not mention IPD sharing.